CLINICAL TRIAL: NCT06077513
Title: Human Alveolar Bone Augmentation: Comparison 3-D CAD-CAM Ti-mesh Frame With a Conventional Ti-Mesh Frame Fabricated at Time of Surgery
Brief Title: Ti-Mesh Frame Comparison for Alveolar Bone Augmentation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-43856; AP 37 (Other: Geistlich Pharma North America Inc)
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Tooth Loss
Keywords: Conventional Ti-Mesh frame; CAD-CAM printed ti-Mesh frame; Dental implants; 3-D Alveolar Bone Augmentation; Surgery time; Post op mesh exposure; Post op bone added
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD-CAM Ti-Mesh frame (Experimental): Participants randomized into this arm will have their tooth loss treated with CAD-CAM designed and preprinted Ti-MESH during surgery.
  Interventions: Procedure: CAD-CAM designed and preprinted Ti-Mesh frame
- Conventional Ti-Mesh frame (Active Comparator): Participants randomized into this arm will have their tooth loss treated with conventional chairside fabrication of Ti-MESH during surgery.
  Interventions: Procedure: Conventional chairside fabrication of Ti-Mesh frame

INTERVENTIONS:
Procedure: CAD-CAM designed and preprinted Ti-Mesh frame — CAD-CAM technology which is the process of designing and manufacturing a custom-made dental device, or a patient-specific dental device from an industrialized product, with the aid of a computer.will be used to plan and preprint a 3-D Ti-Mesh frame prior to the surgery.
  Arms: CAD-CAM Ti-Mesh frame
Procedure: Conventional chairside fabrication of Ti-Mesh frame — A three-dimensional frame or cage of Ti-Mesh or Ti-reinforced d-polytetrafluoroethylene (PTFE) will be fashioned during the surgery to contain, shape and stabilize the bone graft materials (the internal scaffold). This 3-D frame will be custom fabricated from a perforated Ti Mesh sheet material at the time of surgery which takes considerable time and skill.
  Arms: Conventional Ti-Mesh frame

SUMMARY:
This research compares a chairside Titanium Mesh frame fabrication used during bone grafting procedures with the use of a computer-aided design/computer-assisted manufacture (CAD-CAM) Titanium Mesh frame. In addition, a novel method of measuring soft tissue thickness will be tested using an Optical scanner at various times during the sequence of surgeries.

The device used for shaping is a very thin, perforated titanium metal sheet with numerous small perforations (referred to as Micromesh). The construction of this device is usually accomplished chairside at the time of the surgery with custom cutting and shaping done using cues from the geometry of the surgical defect. An alternative approach will be tested where the mesh is pre-designed using digital information provided by a special xray and an optical scan device which takes a digital impression of the tooth and soft tissue surface. A digitally designed frame can then be printed using CAD-CAM software prior to surgery. This should reduce surgical time.

A randomized control trial of 30 patients needing 3-D bone augmentation will be conducted comparing chairside fabrication of Ti-MESH or TEST- CAD-CAM designed and preprinted Ti-MESH to investigate these objectives:

1. Compare the operative times required for placement and removal of two different Ti-MESH frame fabrications
2. Compare post-op wound healing -Ti MESH exposure rates, bone production (volume, contour, and quality) and soft tissue thickness changes during the 1-year study period.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous
* Adult dental patients that require moderate 3-D bone augmentation for dental implant site improvement

Exclusion Criteria:

* Poor oral hygiene indices for microbial plaque (PI) and gingival inflammation (GI)
* Patients who have been on Chemotherapy or Radiation therapy within last 5 years.
* Patients under active treatment with following medications: Bisphosphonates, Gabapentin, Glucocorticoids, Methotrexate, or Estrogen supplements.
* Subjects under the direct supervision of the PI
* Smoking more than 10 cigarettes per day
* Uncontrolled diabetes or other metabolic disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Bone contour accuracy | 5 months post op
  Bone contour accuracy will be derived by merger of the post op Cone beam computed tomography (CBCT) DICOM file with the CBCT-1/CEREC-1/Virtual Implant file produced at the planning stage. Accuracy of fit will be calculated for volume and linear measures (4 sides of each implant-MDBL) horizontal and vertical from the implant restorative platform.
Total surgical time | 2 hours
  Total surgical time is defined as from incision time to completion of sutures and will be measured in minutes.
Surgical exposure time for recipient site | 5 minutes
  Surgical exposure time will be measured for recipient site in minutes

SECONDARY OUTCOMES:
Ti-Mesh exposure incidence | 1 week, 2 weeks, 4weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks
  Number of exposures
Ti-Mesh exposure size | 1 week, 2 weeks, 4weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks
  Ti-Mesh exposure size will be measured in millimeters
Ti-Mesh exposure location | 1 week, 2 weeks, 4weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks
  Ti-Mesh exposure location will be documented within mucosa, gingiva, or at the incision line
Percentage of Vital bone | 6 months
  Percentage of vital bone will be measured in histologic sections of bone core taken at time of implant surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Serge Dibart, DMD, Principal Investigator — BU Goldman School of Dental Medicine, Oral Biology/Periodontics; Albert M Price, DMD, Study Director — BU Goldman School of Dental Medicine, Oral Biology/Periodontics
Locations (1):
- BU Goldman School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No